CLINICAL TRIAL: NCT03353740
Title: Gallium-68 PSMA-11 PET Imaging in Patients With Biochemical Recurrence
Brief Title: Gallium-68 PSMA-11 Positron Emission Tomography (PET) Imaging in Patients With Biochemical Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 175518; NCI-2018-00040 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 labeled PSMA-11 PET (Experimental): PSMA PET imaging: Patients will receive Ga-68 labeled PSMA-11 PET and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled PSMA-11 PET

INTERVENTIONS:
Drug: Ga-68 labeled PSMA-11 PET — Patients will be imaged using Ga-68 labeled PSMA-11 PET to determine if the presence of metastatic disease. Prostate Specific Membrane Antigen (PSMA) is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protocol.
  Other Names: Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled Glu-NH-CO-NH- Lys(Ahx)-HBED-CC; Ga-68 labeled Glu-urea- Lys(Ahx)-HBED-CC; Ga-68 labeled HBED-CC PSMA

SUMMARY:
The investigators are imaging patients with prostate cancer using a new PET imaging agent (Ga-68-PSMA-11) in order to evaluate its ability to detection prostate cancer in patients with biochemical recurrence after prostatectomy and radiation therapy.

ELIGIBILITY:
Inclusion Criteria

* Histopathologically proven prostate adenocarcinoma.
* Rising prostate-specific antigen (PSA) (at least two consecutive rising PSAs) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

  * Post radical prostatectomy (RP) - American Urological Association (AUA) recommendation for biochemical recurrence after radical prostatectomy

    * PSA greater than or equal to 0.2 ng/mL measured more than 6 weeks after RP.
  * Post-radiation therapy -ASTRO-Phoenix consensus definition of biochemical recurrence after radiation therapy

    * Nadir + greater than or equal to 2 ng/mL rise in PSA
* Karnofsky performance status of > 50 (or Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) equivalent).
* Age >= 18.
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria

* Unable to lie flat, still or tolerate a PET scan.
* Concomitant investigational therapy.
* Patient undergoing active treatment for non-prostate malignancy, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.
* Contraindication to furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. (Note: This exclusion criteria can be removed if Furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction is available for the used PET device).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets were made available to collaborating researchers
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Fendler WP, Calais J, Eiber M, Simko JP, Kurhanewicz J, Santos RD, Feng FY, Reiter RE, Rettig MB, Nickols NG, Kishan AU; PSMA PET Reader Group; Slavik R, Carroll PR, Lawhn-Heath C, Herrmann K, Czernin J, Hope TA. False positive PSMA PET for tumor remnants in the irradiated prostate and other interpretation pitfalls in a prospective multi-center trial. Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):501-508. doi: 10.1007/s00259-020-04945-1. Epub 2020 Aug 17. PMID 32808077
- [Derived] Fendler WP, Calais J, Eiber M, Flavell RR, Mishoe A, Feng FY, Nguyen HG, Reiter RE, Rettig MB, Okamoto S, Emmett L, Zacho HD, Ilhan H, Wetter A, Rischpler C, Schoder H, Burger IA, Gartmann J, Smith R, Small EJ, Slavik R, Carroll PR, Herrmann K, Czernin J, Hope TA. Assessment of 68Ga-PSMA-11 PET Accuracy in Localizing Recurrent Prostate Cancer: A Prospective Single-Arm Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):856-863. doi: 10.1001/jamaoncol.2019.0096. PMID 30920593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ga-68 Labeled PSMA-11 PET
Started | 346
Completed | 294
Not Completed | 52
Not completed — Images for these participants not viable | 52

BASELINE CHARACTERISTICS:
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 346
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 2
  50-59 years old | 22
  60-69 years old | 125
  70-79 years old | 157
  80-89 years old | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 346
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 323
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 7
  White | 276
  More than one race | 1
  Unknown or Not Reported | 40
Region of Enrollment [Number; unit: participants]
  United States | 346

OUTCOME MEASURES:

1. Primary Outcome: True Positive Rate for Detection of Tumor Location in Lymph Nodes Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the lymph nodes using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. Corresponding two-sided 95% confidence intervals will be constructed using the Wilson score method.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

2. Primary Outcome: True Positive Rate for Detection of Tumor Location in Visceral Tissue Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the visceral tissue using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. Corresponding two-sided 95% confidence intervals will be constructed using the Wilson score method.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

3. Primary Outcome: True Positive Rate for Detection of Tumor Location in Bone Tissue Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the bone tissue using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. Corresponding two-sided 95% confidence intervals will be constructed using the Wilson score method.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

4. Primary Outcome: True Positive Rate for Detection of Tumor Location in Prostate Bed Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the prostate bed using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy, clinical and conventional imaging follow-up. Corresponding two-sided 95% confidence intervals will be constructed using the Wilson score method.
Time Frame: 1 day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

5. Secondary Outcome: Positive Predictive Value (PPV) for Detection of Tumor Location in Lymph Nodes Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up.
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the lymph nodes as confirmed by by histopathology/biopsy, clinical and conventional imaging follow-up.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

6. Secondary Outcome: PPV for Detection of Tumor Location in Visceral Lesions Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up.
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in visceral tissue as confirmed by by histopathology/biopsy, clinical and conventional imaging follow-up.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

7. Secondary Outcome: PPV for Detection of Tumor Location in Bone Metastasis Lesions Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up.
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer metastasized in the bone as confirmed by by histopathology/biopsy, clinical and conventional imaging follow-up.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

8. Secondary Outcome: PPV for Detection of Tumor Location in Prostate Bed Confirmed by Histopathology/Biopsy, Clinical and Conventional Imaging Follow-up.
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the prostate bed as confirmed by by histopathology/biopsy, clinical and conventional imaging follow-up.
Time Frame: 1 Day
Population: Data on clinical and conventional imaging follow-up not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

9. Secondary Outcome: True Positive Rate for Detection of Tumor Location in Lymph Nodes Confirmed by Histology/Pathology Only
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the lymph nodes using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy only.
Time Frame: 1 Day
Population: Only 7 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 7
proportion of participants | 0.40

10. Secondary Outcome: True Positive Rate for Detection of Tumor Location in Visceral Tissue Confirmed by Histology/Pathology Only
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the visceral tissue using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy only.
Time Frame: 1 Day
Population: Only 9 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 9
proportion of participants | 0.86

11. Secondary Outcome: True Positive Rate for Detection of Tumor Location in Bone Tissue Confirmed by Histology/Pathology Only
Description: The true positive rate or detection rate (sensitivity) is defined as the proportion of all participants who have prostate cancer detected in the bone tissue using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy only.
Time Frame: 1 Day
Population: Only 2 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 2
proportion of participants | 1.00

12. Secondary Outcome: True Positive Rate for Detection of Tumor Location in Prostate Bed Confirmed by Histology/Pathology Only
Description: The true positive rate or detection rate is defined as the proportion of all participants who have prostate cancer detected in the prostate bed using Ga68-PSMA-11, where disease location is also confirmed by histopathology/biopsy only.
Time Frame: 1 Day
Population: Only 30 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 30
proportion of participants | 0.88

13. Secondary Outcome: PPV for Detection of Tumor Location in Lymph Nodes Confirmed by Histopathology/Biopsy Only
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the lymph nodes as confirmed by by histopathology/biopsy
Time Frame: 1 Day
Population: Only 7 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 7
proportion | 0.5

14. Secondary Outcome: PPV for Detection of Tumor Location in Visceral Tissue Confirmed by Histopathology/Biopsy Only
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the visceral tissue as confirmed by by histopathology/biopsy
Time Frame: 1 Day
Population: Only 9 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 9
proportion | 0.86

15. Secondary Outcome: PPV for Detection of Tumor Location in Bone Tissue Confirmed by Histopathology/Biopsy Only
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the bone tissue as confirmed by by histopathology/biopsy
Time Frame: 1 Day
Population: Only 2 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 2
proportion | 1.00

16. Secondary Outcome: PPV for Detection of Tumor Location in Prostate Bed Confirmed by Histopathology/Biopsy Only
Description: Positive predictive value is the probability that participants with a positive reading truly have prostate cancer in the prostate bed as confirmed by by histopathology/biopsy
Time Frame: 1 Day
Population: Only 30 participants had adequate histology/biopsy data for this analysis
Measure: Number; unit: proportion
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 30
proportion | 0.92

17. Secondary Outcome: Detection Rate of 68Ga-PSMA-11 PET Stratified by Prostate-specific Antigen (PSA) Value
Description: Detection rate (sensitivity) on a per-patient basis of 68Ga-PSMA-11 PET stratified by PSA value (0.2- <0.5, 0.5 - <1.0, 1.0 - <2.0, 2.0 - <5.0, >=5.0) will be summarized in tabular format for participants with PSMA positive disease, independent of pathology, imaging or clinical follow-up.
Time Frame: 1 Day
Population: The number analyzed per row represents the number of participants in each category
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 294
proportion of participants
  PSA = < 0.5: number analyzed (Participants) | 55
  PSA = < 0.5 | 0.53
  PSA = 0.5 - <1.0: number analyzed (Participants) | 38
  PSA = 0.5 - <1.0 | 0.68
  PSA = 1.0 - <2.0: number analyzed (Participants) | 38
  PSA = 1.0 - <2.0 | 0.68
  PSA = 2.0 - <5.0: number analyzed (Participants) | 82
  PSA = 2.0 - <5.0 | 0.93
  PSA >= 5.0: number analyzed (Participants) | 81
  PSA >= 5.0 | 0.94

18. Secondary Outcome: Detection Rate of 68Ga-PSMA-11 PET Stratified by Prior Cancer Treatment
Description: Detection rates (sensitivity) on a per-patient basis of 68Ga-PSMA-11 PET stratified by prior cancer treatment (Prostatectomy, Radiation, or Prostatectomy plus Radiation) will be summarized in tabular format.
Time Frame: 1 Day
Population: Prior cancer treatment for only 287 evaluable participants was collected. The number analyzed per row represents the number of participants in each category.
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 287
proportion of participants
  Prostatectomy only: number analyzed (Participants) | 87
  Prostatectomy only | 0.93
  Radiation therapy only: number analyzed (Participants) | 110
  Radiation therapy only | 0.65
  Prostatectomy and salvage radiation therapy: number analyzed (Participants) | 90
  Prostatectomy and salvage radiation therapy | 0.84

19. Secondary Outcome: Detection Rate of 68Ga-PSMA-11 PET Stratified by Prior Use of Androgen Deprivation Therapy (ADT)
Description: Detection rate (sensitivity) on a per-patient basis of 68Ga-PSMA-11 PET stratified by prior use of ADT as a cancer treatment (Prior treatment with ADT, No prior treatment with ADT) will be summarized in tabular format.
Time Frame: 1 Day
Population: Prior ADT treatment for only 272 evaluable participants was collected. The number analyzed per row represents the number of participants in each category.
Measure: Number; unit: proportion of participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 272
proportion of participants
  Prior treatment with ADT: number analyzed (Participants) | 15
  Prior treatment with ADT | 0.8
  No prior treatment with ADT: number analyzed (Participants) | 257
  No prior treatment with ADT | 0.8

20. Secondary Outcome: Percent of Participants With a Change in Clinical Management
Description: Impact of 68Ga-PSMA-11 PET on clinical management in patients with biochemical recurrence (BCR) was measured using Pre-PET (Q1), post-PET (Q2), and post-treatment (Q3) questionnaires sent to referring physicians recording site of recurrence and intended (Q1 to Q2 change) and implemented (Q3) therapeutic and diagnostic management. Percentage of participants with a change in clinical management will be reported using descriptive statistics based on qualitative physician responses from the change in management surveys.
Time Frame: Up to 6 months
Population: Data on change in clinical management not collected for this sample
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

21. Secondary Outcome: Rate of Inter-reader Reproducibility for Positivity
Description: Inter-reader reproducibility for positivity at the patient level will be reported using the Fleiss' Kappa test for multiple readers
Time Frame: 1 Day
Population: Inter-reader reproducibility data not collected
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 0

22. Secondary Outcome: Number of Participants With Grade 3 or Higher, Treatment-related Adverse Events
Description: All grade 3 and above adverse events will be recorded using the NCI CTCAE v4.0. The Investigator will assign attribution of the possible association of the event with use of the investigational drug.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ga-68 Labeled PSMA-11 PET
Number analyzed (Participants) | 346
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Ga-68 Labeled PSMA-11 PET
All-Cause Mortality (participants affected / at risk) | 0/346
Serious Adverse Events (participants affected / at risk) | 0/346
Other Adverse Events (participants affected / at risk) | 0/346

LIMITATIONS AND CAVEATS:
Only a small sample of participants had viable tissue for histological confirmation outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT03353740/Prot_SAP_000.pdf